CLINICAL TRIAL: NCT01144169
Title: A Phase IB Study of Hydroxychloroquine Prior to Nephrectomy in Patients With Primary Renal Cell Carcinoma
Brief Title: Study of Hydroxychloroquine Before Surgery in Patients With Primary Renal Cell Carcinoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: barriers to accrual: delay until surgery and additional pre-operative visits
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Jodi Maranchie, MD, FACS, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-029
Record Dates: First submitted 2010-06-10; First posted 2010-06-15 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Renal Cell Carcinoma
Keywords: Renal cell carcinoma; Hydroxychloroquine; Nephrectomy; Autophagy
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hydroxychloroquine (HC) (Experimental): HC orally for 14 days prior to nephrectomy
  Interventions: Drug: Hydroxychloroquine (HC)

INTERVENTIONS:
Drug: Hydroxychloroquine (HC) — Subjects will receive HC orally for 14 days prior to surgery. The fixed dose of HC will be 400 mg/day in divided doses (200 mg bid). The final dose will be administered on the evening prior to nephrectomy.
  Other Names: Plaquenil®

SUMMARY:
The main goal of this research study is to determine whether treating patients with renal cell cancer with hydroxychloroquine before surgery can make the cancer easier to kill. Another goal is to see how the study drug affects the body's immune cells which fight cancer cells.

DETAILED DESCRIPTION:
Autophagy is a cellular survival mechanism that protects from stress-induced programmed death. Autophagy may enable renal cancer to escape from cytokine therapy, cytotoxic chemotherapy or targeted agents. Hydroxychloroquine prevents autophagy by blocking acidification of lysosomes, and is being studied in clinical trials as a means of enhancing of cancer therapy. This phase Ib clinical trial will test the hypothesis that pre-operative exposure to HC reduces biologic markers of autophagy in peripheral blood, normal kidney and renal cancer specimens obtained at the time of nephrectomy. These data will be used in the design and pharmacodynamic monitoring of future therapeutic trials of HC in combination with high dose interleukin-2 and other systemic therapies for advanced RCC.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with suspected primary or metastatic RCC (stage 1-IV) with planned nephrectomy or partial nephrectomy.
* ECOG performance status ≤1
* Normal renal, hepatic, and hematologic function at the time of enrollment as evidenced by:

  * Serum creatinine level ≤1.5 the upper limits of normal (ULN)
  * Serum total bilirubin level ≤1.5 X ULN
* White blood cell count > or = 3.5x109/ml per ml and platelet count ≥ 100x109 per ml
* Age >18 years.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Subjects who have received chemotherapy for any diagnosis within 12 months prior to study entry.
* Prior use of radiotherapy or investigational agents for RCC.
* Concurrent malignancies with evidence of active or measurable disease except non-melanoma skin cancer
* Inability to adhere to study and/or follow-up procedures
* History of allergic reactions or hypersensitivity to the study drug (hydroxychloroquine) or current therapy with the study drug for other reasons.
* Other concurrent experimental therapy.
* The effects of HC on the developing human fetus are unknown. For this reason women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. All females of childbearing potential must have a blood test or urine study within two weeks prior to registration to rule out pregnancy. Should a woman become pregnant while participating in this study, she should inform her treating physician immediately. If a man impregnates a woman while participating in this study, he should inform his treating physician immediately as well.
* HIV-positive patients are not excluded from the study. However, for patients receiving combination anti-retroviral therapy, the potential impact of pharmacokinetic interactions with HC is unknown. Therefore, HIV-positive patients actively receiving anti-retroviral therapy are excluded from the study.
* Patients with psoriasis are ineligible unless the disease is well controlled and they are under the care of a specialist who agrees to monitor the patient for exacerbations.
* Patients requiring the use of enzyme-inducing anti-epileptic medication that includes: phenytoin, carbamazepine, phenobarbital, primidone or oxcarbazepine are excluded. Hydroxychloroquine is known to affect the CYP2D6 metabolic pathway. A list of drugs with potential interaction is included in Appendix H.
* Patients with previously documented macular degeneration or diabetic retinopathy are excluded.
* Patients with known glucose-6-phosphate dehydrogenase (GP6D) deficiency
* EKG with QTc >500 msec at baseline (average of 3 determinations at 10 minutes interval). Subjects with ventricular pacemaker for whom QT interval is not measurable will be eligible on a case-by-case basis.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-10; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Measure biologic markers of autophagy in tumor and normal tissues (peripheral blood mononuclear cells, renal parenchyma) following a short course of pre-operative oral hydroxychloroquine [HC] in patients with renal cell carcinoma. | Pre-hydroxychloroquine (HC), post-HC/pre-nephrectomy, post-nephrectomy (up to 1 month)

SECONDARY OUTCOMES:
Measure the serum biomarker response (HMGB1, sRAGE, VEGF, fibronectin, CRP, IL-6, nicotinamide N-methyltransferase, thrombospondin-1, CD 14, and ferritin) following pre-operative oral HC. | One month post-nephrectomy
Assess the effect of pre-operative HC on phenotype and function of DC and NK cells | One month post-nephrectomy
Assess the effect of pre-operative HC on abundance of neutrophils, NK cells, T-cells and T-cell subsets, PDCs and MDCs in the resected tumor, expression of CAIX and NOX4 compared with matched age/sex/histology matched controls. | One month post-nephrectomy
Assess miRNAs pre and post HC and postoperatively in blood and in resected tumor and normal kidney compared to stage- and grade-matched controls. | Pre-HC, post-HC/pre-nephrectomy, post-nephrectomy (1 month)

CONTACTS AND LOCATIONS:
Overall Officials: Jodi K. Maranchie, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (2):
- United States (2):
  - UPCI/UPMC Cancer Centers, Pittsburgh, Pennsylvania
  - UPMC Department of Urology, Pittsburgh, Pennsylvania